CLINICAL TRIAL: NCT00059293
Title: TCD Ultrasound of Subjects Enrolled in Baby Hug (Baby TCD)
Brief Title: Transcranial Doppler (TCD) Ultrasound of Subjects Enrolled in BABY HUG - Ancillary to BABY HUG
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1208; R01HL072946 (NIH)
Record Dates: First submitted 2003-04-22; First posted 2003-04-24 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2008-07

CONDITIONS: Blood Disease; Anemia, Sickle Cell; Cerebrovascular Disorders; Cerebral Embolism and Thrombosis
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell; Cerebrovascular Disorders; Intracranial Embolism and Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To use transcranial Doppler (TCD) ultrasound to detect stroke risk in children with sickle cell disease.

DETAILED DESCRIPTION:
BACKGROUND:

Cerebral vasculopathy and stroke are among the most serious complications of sickle cell disease. Not every patient will develop central nervous system disease but most children have some evidence of cognitive impairment and about 10% will have overt stroke if this is not forestalled by transcranial Doppler (TCD) screening, identification of individuals at greatest risk by estimating maximal cerebral blood flow and commencing prophylactic transfusion. The basis of these recommendations is studies in children over age 2-years where stroke is most prevalent. Transfusion is not without its own serious and considerable risks so that other measures for delaying or preventing cerebral vasculopathy would be valuable. Hydroxyurea (HU) can reduce both morbidity and mortality of sickle cell anemia in adults; most likely the same pertains in children. Unknown are the effects of HU in infants and the youngest children and whether its successful use can reduce the risks of sickle cerebrovascular disease. If HU is associated with reduced TCD velocity, and if it is safe in infants, the medical implications would be high.

Baby TCD is an ancillary study to the initial phase of BABY HUG, a multicenter clinical trial funded by the NHLBI. In BABY HUG, infants (12-17 months old) with sickle cell disease (SCD) will be randomized to either hydroxyurea (HU) or placebo and followed for 24 months. There is broad interest in the effect of hydroxyurea on the central nervous system in the children being studied. Stroke occurs after age 1 year and there is evidence that the process of cerebrovascular disease starts very early in some patients. The Cooperative Study of Sickle Cell Disease documented a high risk of incident stroke in the 2-6 year age group. The study is in response to an initiative on Ancillary Studies in Heart, Lung, and Blood Disease Trials released in June, 2000.

DESIGN NARRATIVE:

The study will perform TCD on the 40 children in BABY HUG at baseline and at the end of study. TCD has proven very useful in estimation of stroke risk in children with SCD ages 2-16 years, and is at the center of a paradigm of primary stroke prevention recommended by the National Heart, Lung, and Blood Institute based on the STOP study. If stroke risk could be detected at an earlier stage (i.e., younger than the 2-16 year-old subjects in STOP), then physicians would be able to provide preventive treatment at an earlier stage of the disease. TCD will be performed before and after 24 months of treatment. TCD performance and reading will be centrally controlled and STOP-consistent. The investigators have experience in TCD of infants, the age targeted by the parent study. TCD will be compared between HU and control groups, before and after treatment. In addition, the investigators have access to data from over 400 children in the 2-4 year age range from the STOP screening program performed in the mid- to late 1990s. Since these patients were not on HU or transfusion this dataset will be used to give an estimate of the prevalence of high stroke risk without HU treatment, and can be compared to the HU group in Baby HUG, adding another important comparative dimension to the analyses. Although the sample size is purposely small as designed by the parent study, large differences in the prevalence of high-risk patients at the end of treatment could be detected by Baby TCD.

ELIGIBILITY:
No eligibility criteria

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The BABY HUG Follow-up Study I was an observational study to provide structured monitoring of the subjects enrolled in the BABY HUG Treatment Study, to initiate characterization of the long-term toxicities and unexpected risks (if any) associated with treatment with hydroxyurea at an early age, and any potential benefits of therapy.
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams, Principal Investigator — Medical University of South Carolina